CLINICAL TRIAL: NCT05399095
Title: Supine Positioning for Graft Attachment After Descemet Membrane Endothelial Keratoplasty: a Randomized Controlled Trial
Brief Title: Supine Positioning for Graft Attachment After Descemet Membrane Endothelial Keratoplasty
Acronym: SUPER-DMEK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Eye Hospital, Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETK 22-1101
Record Dates: First submitted 2022-05-22; First posted 2022-06-01 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Fuchs' Endothelial Dystrophy
Keywords: Fuchs' endothelial corneal dystrophy; Descemet membrane endothelial keratoplasty; Incomplete graft attachment; Endothelial corneal graft detachment; Rebubbling (repeat injection of air or gas in the anterior chamber); Supine positioning; Postoperative posture; Anterior segment optical coherence tomography; Neural network; Machine learning; Randomized controlled trial
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Intervention Model Description: Stratification will be performed according to the surgical procedure (DMEK alone or DMEK combined cataract surgery). Within each strata, participants will be randomized in a 1:1 ratio to 5 days (intervention) and 1 day (control) postoperative supine positioning.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, surgeons, and investigators will be masked until the first postoperative day after DMEK. Investigators will open the opaque envelope with the study assignment together with the participant and inform care providers on the positioning regimen for the next 4 days.
  The primary outcome will be assessed by a masked investigator using a trained and validated neural network for image segmentation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 days supine positioning (Experimental): Supine positioning for 5 days after DMEK with upright positioning for only 10 min every hour.
  Interventions: Behavioral: Supine positioning: 5 days
- 1 day supine positioning followed by usual physical activity for 4 days (Active Comparator): Supine positioning for 1 days after DMEK with upright positioning for only 10 min every hour.
  Interventions: Behavioral: Supine positioning: 1 days

INTERVENTIONS:
Behavioral: Supine positioning: 5 days — Supine positioning for 5 days after DMEK
  Arms: 5 days supine positioning
Behavioral: Supine positioning: 1 days — Supine positioning for 1 days after DMEK
  Arms: 1 day supine positioning followed by usual physical activity for 4 days

SUMMARY:
This randomized controlled trial evaluates the efficacy and safety of postoperative supine head positioning on graft attachment after Descemet membrane endothelial keratoplasty in patients with Fuchs' endothelial corneal dystrophy (FECD).

DETAILED DESCRIPTION:
In Descemet membrane endothelial keratoplasty (DMEK), an air or gas bubble is inserted in the anterior chamber of the eye to keep the ultrathin endothelial corneal graft attached to the patients own cornea. Supine positioning is thought to improve attachment by using the tamponade effect of the bubble. At present, it is unclear how long supine positioning is required. Positioning regimens vary between one hour to over one week. In this trial, the investigators will assess if prolonged supine positioning for 5 days improves graft attachment and long-term outcomes compared to supine positioning for 1 day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced Fuchs' endothelial corneal dystrophy (FECD)
* Indication for corneal endothelial transplantation (Descemet Membrane Endothelial Keratoplasty - DMEK)

Exclusion Criteria:

* Other corneal diseases (i.e. corneal scars, corneal dystrophies except FECD, corneal inflammation / infection)
* Regular use of drugs potentially affecting the cornea (i.e. amiodarone, chloroquine, triptan, isotretinoin, use of contact lenses in past four weeks, anesthetic eye drops)
* Diabetes mellitus with endorgan complications)
* Lack of fixation during corneal tomography
* Bedridden

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Graft attachment | At two weeks after DMEK
  Area of graft detachment, quantified from a trained and validated neural network for image segmentation of anterior segment optical coherence tomography
Graft attachment | At two weeks after DMEK
  Volume of graft detachment, quantified from a trained and validated neural network for image segmentation of anterior segment optical coherence tomography

SECONDARY OUTCOMES:
Rebubbling | At two weeks and 3 months after DMEK
  Number of eyes with secondary injection of air after DMEK
Safety of supine positioning | At two weeks and 3 months after DMEK
  Adverse events (AE) and serious AEs (SAE)
Subjective visual function | At 3, 12, and 24 months after DMEK
  Subjective visual function on a scale from 0 (worse vision) to 10 (best vision) with higher scores meaning better subjective visual function
Visual acuity | At 3, 12, and 24 months after DMEK
  Best-corrected visual acuity to determine visual acuity in letters
Disability glare | At 3, 12, and 24 months after DMEK
  Straylight meter measurement to determine forward scatter in logs straylight parameter
Graft health: endothelial cell density | At 3, 12, and 24 months after DMEK
  Specular microscopy to determine endothelial cell density
Graft health | At 12, and 24 months after DMEK
  Slit-lamp exam to identify signs of graft rejection
Patient-reported visual disability | At 3, 12, and 24 months after DMEK
  The Visual Acuity Factor and Glare Factor of the Visual Function and Corneal Health Status (V-FUCHS) instrument. The instrument's scores are Rasch-analysis based scores expressed in logits. Participants with more difficulty have higher or more positive V-FUCHS scores.
Corneal edema | At 2 weeks and at 3, 12, and 24 months after DMEK
  Tomography to determine corneal edema in µm
Corneal backscatter | At 3, 12, and 24 months after DMEK
  Tomography to determine corneal backscatter in scatter units (SU)

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Wacker, MD FEBO, Principal Investigator — University of Freiburg, Eye Hospital
Locations (1):
- Medical Center - University of Freiburg, Eye Hospital, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No